CLINICAL TRIAL: NCT01896401
Title: InSeal Vascular Closure Device Clinical Study Protocol
Acronym: VCD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Initiated a new study with improved device
Sponsor: InSeal Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-14-003
Record Dates: First submitted 2013-07-06; First posted 2013-07-11 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Percutaneous Closure of Artery Access Sites
Keywords: large bore endovascular catheterization procedures; Vascular Closure Device

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- InSeal's Vascular Closure Device (Experimental): Use of the experimental VCD to close the access site of the artery
  Interventions: Device: InSeal's Vascular Closure Device

INTERVENTIONS:
Device: InSeal's Vascular Closure Device

SUMMARY:
The InSeal vascular closure device (VCD)is assessed as percutaneous closure of artery access sites for quick hemostasis and ambulation in patients who have undergone large bore endovascular catheterization procedures.

The study hypothesis is that the VCD is safe and efficaient in achieving hemostasis in the study population.

ELIGIBILITY:
Inclusion Criteria:

* Candidate for large bore catheterization procedure (such as TAVI, aortic endograft repair) using a CE approved 18Fr access sheath.
* Subject age is at least 18 years
* Patient has signed most recent approved version of the Informed Consent
* Existence of an additional arterial access port is required in instances where an occluding balloon is planned to be used as a safety precaution.

Exclusion Criteria:

* Women Of Child Bearing Potential (WOCBP)
* Legally non-competent patients
* Patient participating in another clinical study at the time of the InSeal VCD study
* Prior target artery closure with a vascular closure device having intravascular component (such as Angio-Seal) 30 days prior to catheterization
* Subjects with known coagulopathy, preexisting hematoma, arteriovenous fistula, or pseudoaneurysm at the vessel access site prior to artery closure
* Patients that do not tolerate aspirin and clopidogrel anticoagulation treatment
* Prior vascular surgery or vascular graft in region of access site
* Significant calcification, atherosclerotic disease, or stent within 1.5 cm of the puncture site that may interfere with the operation of the experimental device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2012-02; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
1. Hemostasis within 15 minutes following vessel access site closure and after ACT falls below 200 second | 15 minutes

SECONDARY OUTCOMES:
2. Combined rate of closure-device related major adverse events in first month | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Cardio Vascular Centrum Frankfurt, Frankfurt, Germany